CLINICAL TRIAL: NCT06556771
Title: Comparison of Gongs Mobilization and Kaltenborn Mobilization on Mechanical Neck Pain
Brief Title: Comparison of Gongs and Kaltenborn Mobilization on Neck Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Komal Shahzad
Record Dates: First submitted 2024-08-13; First posted 2024-08-16 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Mechanical Neck Pain
Keywords: Gongs mobilization, Kaltenborn mobilization , Mechanical neck pain , proprioception
MeSH Terms: interventions — Traction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Gongs mobilization and conventional therapy , sessions 3 per week , mobilization for 5 minutes and 30 minutes session for total 4 weeks. exercise 3 sets for 10 repetitions.
  Modality (Hydrocollator pack, TENS for 15 minutes with pulse frequency of 10-200 Hz, pulse width 100 - 250 micro seconds.
  Interventions: Other: Gongs mobilization + conventional physical therapy
- Group B (Experimental): Kaltenborn mobilization along with cervical traction and conventional therapy:
  Intervention will be given 3 times/week 5 minutes mobilization Exercise 3 sets for 10 repetitions and 30 minutes session for 4 consecutive weeks.
  Modality including (Hydrocollator pack, TENS for 15 minutes with pulse frequency of 10-200 Hz, pulse width 100 - 250 micro seconds. Intensity tolerated by patients.
  Interventions: Other: Kaltenborn mobilization along with traction + conventional therapy

INTERVENTIONS:
Other: Gongs mobilization + conventional physical therapy — 3 per week , mobilization for 5 minutes , exercise 3 sets for 10 repetitions for 4 consecutive weeks
  Arms: Group A
Other: Kaltenborn mobilization along with traction + conventional therapy — 3 per week , mobilization for 5 minutes , exercise 3 sets for 10 repetitions for 4 consecutive weeks.
  Arms: Group B

SUMMARY:
The aim of this randomized controlled trial is to find the effect of Gongs mobilization in comparison with Kaltenborn mobilization on mechanical neck pain , range of motion and proprioception.A randomized control trial that will include total 44 participants. The first group will receive Gongs mobilization along with conventional therapy and 2nd group will receive Kaltenborn mobilization along with conventional therapy.

DETAILED DESCRIPTION:
: Neck pain is most common problem with point prevalence of almost 13% and lifetime prevalence of approximately 50%. Mechanical neck pain is defined as nonspecific neck pain arising from anywhere in area bounded above by superior nuchal line and below to first thoracic vertebrae tip and laterally to lateral borders of neck and pain increased by neck movement.

Impairment of cervical proprioception is significant issue in individuals with mechanical neck pain leading to disruption in sensorimotor control in neck. These disruptions can effect posture control and balance. Cervical sensorimotor control involves the central processing of sensory inputs, including visual, vestibular, and cervical proprioceptive information. This process leads to the execution of motor programs by cervical muscles, which plays a crucial role in maintaining head posture, balance, and the stability of cervical joints. Disturbances in cervical sensorimotor control, resulting from neck pain, may potentially lead to additional tissue damage, worsen pain through sensitization in both the peripheral and central nervous systems, and promote dysfunctional motion patterns.

According to literature Gongs mobilization which is an end range mobilization technique introduced by Wontae Gong at all. It has significance that movement of the joint facets other than the fixed one are maximally restricted and mobilization is induced using acceleration and gravity. For mechanical neck pain Kaltenborn mobilization also improved symptoms.

Previous studies worked on effectiveness of Kaltenborn mobilization and Gongs mobilization on neck pain. Aim of this study will be to determine which technique is more in improving pain, ROM and proprioception in mechanical neck pain patients. Our study is related to the fact that it will be helpful for future healthcare provider and will have a significant role in health promotion and spread a healthy lifestyle to public.

ELIGIBILITY:
Inclusion Criteria:

Participants falling in this category would be recruited into the study.

* • Age 18 -65 years

  * Both male and female
  * Primary complaint of neck pain with or without radiating to Upper extremity
  * Pain confined to posterior aspect of neck with mechanical characteristics such as symptoms provoked by neck movement, by palpation of cervical muscles and by sustained posture.
  * Subjects who are willing to participate in study.
  * Patients with Mechanical neck pain

Exclusion Criteria:

* Participants falling in this category would be excluded from the study.

  * Bilateral upper extremity symptoms
  * Whiplash injury
  * Trauma or tumor around neck
  * Previous neck surgery
  * Spinal infection
  * Cervical radiculopathy and myelopathy
  * Vascular syndromes

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-08-09 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-01-10 (Estimated)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale NPRS | 4 weeks
  The NPRS is a segmented numeric version of the visual analog scale which is used to assess pain. It scores ranges from 0-10, 0 means No pain and 10 means Severe pain. Patient will be asked to verbally report the pain score.

SECONDARY OUTCOMES:
: Goniometer | 4 weeks
  : It is an instrument that measures the available range of motion at a joint.
Cervical Joint Position Error | 4 weeks
  The patient is sitting 90 cm from the wall, and the starting point (center of target or reference point) of the laser projection is marked. The patient (blindfolded or closed) performs active neck movement and then returns to the starting position as accurately as possible. The final laser position is measured relative to the starting position (distance or angle). The errors are measured after cervical extension and flexion.

CONTACTS AND LOCATIONS:
Overall Officials: Madiha Ali, MS OMPT, Principal Investigator — Riphah International University
Locations (1):
- Alam Hospital Attock, Attock City, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No